CLINICAL TRIAL: NCT04664855
Title: A Trauma-Informed Approach for Positive Youth Development for Montana Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Lauren Davis, Assistant Professor, Montana State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MontanaSUYear2
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Depression, Anxiety; Suicidal Ideation; Stress; Trauma
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicidal Ideation; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Yoga Group (Experimental): 35 freshman students enrolled in a health and wellness/physical education class at a rural Montana high school
  Interventions: Other: Trauma-Informed Yoga
- Control Group (No Yoga Intervention) (No Intervention): 20 freshman students enrolled in a health and wellness/physical education class at a rural Montana high school

INTERVENTIONS:
Other: Trauma-Informed Yoga — 8 weeks of twice weekly trauma-informed yoga for 45 minutes per session
  Arms: Experimental Yoga Group

SUMMARY:
Given the prevalence of suicide and mental health issues in rural Montana, this project is intended to help mitigate stressors that may contribute to poor behavioral and mental health in high school-aged children. The immediate goal is to measure physical and mental health outcomes in adolescents resulting from a trauma-informed yoga intervention designed to foster positive youth development and student success. It builds on feasibility study for year one in which 19 experimental condition participants engaged in an 8-week yoga program.

DETAILED DESCRIPTION:
mental and physical health issues (17). Stressors deriving from low socioeconomic status and/or traumatic childhood experiences such as abuse or neglect are exacerbated by today's educational culture, where mandated practices such as standardized testing and post-graduation plans are cited as primary causes for stress in adolescents' lives (4).

In Montana, the childhood abuse/neglect rate was 8.3 per 1000 children in 2015, which indicates a 56.8% increase from 2014 (16); nationally, in the same year the abuse/neglect rate was 9 per 1000 children (15). Childhood trauma tends to cluster in areas of high poverty; in Livingston Public Schools in rural southwestern Montana, for instance, 52% of students were eligible for free and reduced-price lunch in 2016, which is the same as the national rate (4; 40). In Livingston, 13.2% of residents are listed as living in poverty, which is slightly above the 12.3% national rate (53). These unfortunate but common childhood stressors can result in significant public health issues including poor mental health, suicidality, substance abuse, juvenile offenses, and autoimmune disease (8). Despite Livingston being on par with national childhood poverty and abuse trends, the suicide rates in Livingston are triple the national average (42). Substance abuse among minors in Montana, which is often comorbid with mental health issues and suicidality, is prevalent; according to a 2015 report by the office of adolescent health, 38% of Montana high schoolers reported having used marijuana at least once, 20% self-reported using alcohol before age 13, and 30% reported using e-cigarettes (36).

Given the prevalence of suicide and mental health issues in rural Montana, this project is intended to cultivate positive coping skills to buffer the negative effects of stressors among school-aged children. Because of the geographic isolation and resulting lack of resources for many schools in Montana, there is a need for innovative and novel school- and community-centered interventions in order to address the varied health needs of rural adolescents. According to research, yoga and mindfulness can have a positive impact on youth development (6; 7; 13; 14). The second year of this pilot study prepares the way for a robust intervention by examining efficacy of this intervention modality compared to a control group in a collaborative school setting, basing the framework of the study on the tenets of community-based participatory research (16). Existing validated measures of efficacy using physical and mental health measures will be used to generate student, teacher, and parent reports of perceived strengths and difficulties, along with measures of anxiety and depressive symptomology. Secondary outcomes of school performance also will be assessed. Efficacy of the intervention will be ascertained through observational and qualitative data obtained utilizing participant, school, and community partner interviews; quantitative feedback will also be gathered from community and school stakeholders to evaluate program outcomes. From this data analysis, decisions regarding any necessary modifications to experimental design and program implementation will be made for third year of the study, which will lead to an expansion to middle level students within the same school district.

Aim 1: Pilot test a trauma-informed yoga intervention for 15-18 year-old male and female high school students.

H1: Students who participate in the pilot intervention will demonstrate improved mental health as measured by a decrease in depressive and anxiety symptomology at the conclusion of the study (week 8) as compared to participants in the control group.

H2: Students who participate in the pilot intervention will demonstrate improved physical health as measured by a decreased resting heart rate, improved sleep patterns, and reduced cortisol levels at the conclusion of the study (week 8) as compared to participants in the control group.

Aim 2: Evaluate the study's school-community-academic partnership at the conclusion of the program using a mixed methods survey. The CAB will meet monthly to determine program adjustments. Survey administration and data analysis will occur in summer 2021. The PI will share results with the CAB to determine areas for program refinement and assess need for study continuation or expansion into multiple schools for year 3.

H3: Findings from the partnership evaluation will be used to refine the community engagement component of the study in Year 3.

This data will be used to determine intervention and program efficacy in order to indicate areas for revision and refinement in year 3 of this study; the data will also inform future implementation plans for program expansion to the middle school level within the same school district.

ELIGIBILITY:
Inclusion Criteria:

Freshmen enrolled in a health and wellness/physical education class at a rural Montana High School

Exclusion Criteria:

None

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Davis, Ed. D, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis L, Aylward A. Mitigating Rural Adolescent Trauma: Remote Delivery of a Trauma-Informed Yoga Intervention During COVID-19. J Child Adolesc Trauma. 2022 Dec 1;16(3):1-14. doi: 10.1007/s40653-022-00496-9. Online ahead of print. PMID 36471891

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Yoga Group: 23 freshman students enrolled in a health and wellness/physical education class at a rural Montana high school
  Trauma-Informed Yoga: 6 weeks of twice weekly trauma-informed yoga for 45 minutes per session
- Control Group (No Yoga Intervention): 22 freshman-senior high school students enrolled in a health and wellness/physical education class at a rural Montana high school
Period: Overall Study
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention)
Started | 23 | 24
Completed | 23 | 22
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The number of intended participants did not volunteer to meet our projected numbers from the initial participant flow section.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention) | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 22 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (0.5) | 16.5 (1.12) | 15.4 (1.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 19
  Male | 7 | 19 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Salivary Cortisol Levels
Description: Students will provide a saliva sample in which cortisol levels will be analyzed through salivary assay kits (through Salimetrics.com). Samples will be collected on the first day of the intervention, halfway through the intervention, and on the last day of the intervention to determine if the intervention has changed cortisol levels. A biostatistician will provide analysis and conclusion of these samples at the conclusion of the study; the mean change pre vs. post is provided here. Negative change indicates improvement in stress levels.
Time Frame: Week 1 and. Week 6
Population: High school students enrolled in a physical education classroom in rural Montana
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention)
Number analyzed (Participants) | 23 | 22
ug/dl | -0.26 (.12) | -0.17 (.27)

2. Secondary Outcome: Patient Health Questionnaire for Adolescents
Description: This 9 item questionnaire is designed to evaluate severity of depressive symptoms in adolescents. It is scored on a Likert scale from 0 (not at all) to 3 (nearly every day) on items linked to depression indicators. The minimum score is a 0 and the maximum score is a 27, and a negative change in score from pre- to post-assessment indicates an improvement in symptomology. Pre and post-intervention means are reported here.
Time Frame: Baseline and 6 weeks
Population: High school students enrolled in a physical education class in rural Montana
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention)
Number analyzed (Participants) | 23 | 22
score on a scale
  Baseline Mean | 8.00 (6.75) | 5.36 (4.89)
  Post-Intervention Mean | 6.39 (6.73) | 4.18 (5.24)

3. Secondary Outcome: Generalized Anxiety Disorder-7 Anxiety Scale
Description: This 7 item questionnaire is based on a Likert scale of 0 (not at all) to 3 (nearly every day) for items related to anxiety disorders. The lowest score is a zero and the maximum score is a 21. A negative change in score from pre- to post-assessment indicates an improvement in symptomology. Pre and post-intervention means are reported here.
Time Frame: Baseline and 6 weeks
Population: High school students enrolled in a physical education class in rural Montana
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention)
Number analyzed (Participants) | 23 | 22
score on a scale
  Pre-Intervention Mean | 6.83 (5.25) | 5.27 (5.13)
  Post-Intervention Mean | 5.35 (5.97) | 4.55 (4.54)

4. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: The CD-RISC 10 is a unidimensional self-reported scale consisting of 10-items measuring resilience. Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4. Possible scores range from 0-100. A higher score indicates higher resilience. Pre and post-intervention means are reported here.
Time Frame: Baseline and 6 weeks
Population: High school students enrolled in a physical education class in rural Montana
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention)
Number analyzed (Participants) | 23 | 22
score on a scale
  Pre-intervention mean | 25.39 (7.45) | 28.32 (7.11)
  Post-Intervention Mean | 24.87 (9.71) | 30.45 (6.44)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Experimental Yoga Group | Control Group (No Yoga Intervention)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04664855/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT04664855/ICF_001.pdf